CLINICAL TRIAL: NCT05926271
Title: POPular GUILTY PILOT: Genotype-guided Clopidogrel Monotherapy
Acronym: POPular GUILTY
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: St. Antonius Hospital (Other)
Responsible Party: Principal Investigator, Jurriën M. ten Berg, MD, PhD, Prof. dr. J.M. ten Berg, St. Antonius Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: NL82555.100.22
Record Dates: First submitted 2023-06-07; First posted 2023-07-03 (Actual); Last update posted 2024-12-03 (Actual); Status verified 2024-11

CONDITIONS: Acute Coronary Syndrome; CYP2C19 Polymorphism
Keywords: Acute coronary syndrome; Monotherapy; P2Y12 inhibitor; Aspirin free strategy
MeSH Terms: conditions — Acute Coronary Syndrome | interventions — Clopidogrel

STUDY DESIGN:
Intervention Model Description: This pilot, genotype-guided clinical trial aims to assess the safety and efficacy of clopidogrel monotherapy in Non-ST-Segment Elevation Acute Coronary Syndrome (NSTE-ACS) patients post-successful percutaneous coronary intervention (PCI). Participants, identified as extensive or ultra-rapid metabolizers by CYP2C19 genotype, will receive clopidogrel monotherapy. The primary outcomes include the ischemic risk (efficacy) and bleeding risk (safety) during the first six months post-PCI. The trial hypothesizes that genotype-guided clopidogrel monotherapy is safe and efficacious in mitigating bleeding and ischemic complications.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Genotype guided arm (Experimental): In this study arm, patients with Non-ST-Segment Elevation Acute Coronary Syndrome (NSTE-ACS) who are extensive or ultra-rapid metabolizers as per their CYP2C19 genotype and have undergone successful percutaneous coronary intervention (PCI) will receive a genotype-guided monotherapy.
  The intervention will be clopidogrel, a potent P2Y12 inhibitor, administered in accordance with the patient's specific genotype. Clopidogrel following PCI will be given with an initial loading dose (300-600mg orally), followed by a maintenance dose of 75mg daily for a defined period, at least 6 months.
  Interventions: Drug: Clopidogrel

INTERVENTIONS:
Drug: Clopidogrel — See arm description earlier.

SUMMARY:
The goal of this pilot clinical trial is to test the safety and effectiveness of genotype-guided clopidogrel monotherapy in patients presenting with Non-ST-Segment Elevation Acute Coronary Syndrome (NSTE-ACS) who have undergone successful Percutaneous Coronary Intervention (PCI). The main questions it aims to answer are:

* Is genotype-guided clopidogrel monotherapy effective in reducing ischemic risk during the first six months following successful PCI?
* Is genotype-guided clopidogrel monotherapy safe in terms of reducing bleeding risk during the first six months following successful PCI?

Participants will be given genotype-guided clopidogrel monotherapy after their successful PCI procedure and will be monitored for any bleeding or ischemic complications over the next six months.

Researchers will compare these results to the typical outcomes associated with traditional Dual antiplatelet therapy (DAPT) to see if genotype-guided clopidogrel monotherapy provides similar or improved protection from ischemic events, but with fewer bleeding complications.

DETAILED DESCRIPTION:
Rationale: Dual antiplatelet therapy (DAPT) consisting of aspirin and a P2Y12 inhibitor is the cornerstone of treatment in patients receiving coronary stent implantation, reducing the risk of stent thrombosis (ST), myocardial infarction (MI) and stroke. However, the need for aspirin is currently challenged as both technical and pharmaceutical advancements reduced atherothrombotic complications such as ST and MI after percutaneous coronary intervention (PCI) and DAPT is associated with bleeding complications. Single antiplatelet therapy (SAPT) after a 1-3 month period of DAPT demonstrated fewer bleeding complications with a similar level of ischemic complications. In addition, potent P2Y12 inhibitor monotherapy was deemed safe without any ST in a pilot study and is currently being investigated in a randomized controlled clinical trial. Since clopidogrel is equally effective in prevention of ischemic complications to ticagrelor and prasugrel in CYP2C19 extensive or ultra-rapid metabolizers, while causing less bleeding complications, this pilot study will explore the safety of genotype-guided clopidogrel monotherapy in CYP2C19 extensive or ultra-rapid metabolizers presenting with Non-ST-Segment Elevation Acute Coronary Syndrome (NSTE-ACS) undergoing successful PCI.

Hypothesis:

Genotype-guided clopidogrel monotherapy is safe in regards to bleeding and ischemic endpoints in NSTE-ACS patients undergoing successful PCI.

Objective:

1. To assess ischemic risk (i.e. efficacy) of genotype-guided clopidogrel monotherapy during the first 6 months following successful PCI in NSTE-ACS patients.
2. To assess bleeding risk (i.e. safety) of genotype-guided clopidogrel monotherapy during the first 6 months following successful PCI in NSTE-ACS patients.

ELIGIBILITY:
Inclusion Criteria:

Patients aged 18 years or older are eligible for inclusion if all of the following criteria are met:

* Clinical diagnosis of NSTE-ACS (i.e. NSTEMI or unstable angina)
* Successful PCI (according to the treating physician) with implantation of new generation drug eluting stents.
* CYP2C19 extensive or ultra-rapid metabolizer

Exclusion Criteria:

A potential subject who meets any of the following criteria will be excluded from participation in this study:

* CYP2C19 poor or intermediate metabolizer
* Known allergy or contraindication for aspirin or clopidogrel.
* Concurrent use of oral anticoagulants (e.g. because of atrial fibrillation)
* Ongoing indication for DAPT at admission (e.g. due to recent PCI or ACS)
* High-risk features for PCI including left main disease, chronic total occlusion, bifurcation lesion requiring 2-stent treatment, saphenous or arterial graft lesion, severely calcified lesion requiring the use of the Rotablator system, ≥3 treated vessels, ≥ 3 stents implanted and total stent length >60 mm
* Recent stroke, transient ischemic attack (TIA) or intracranial bleeding
* Severe hepatic impairment (Child Pugh class C)
* Planned surgical intervention within 6 months of PCI
* Patients requiring staged procedure (to avoid heterogeneity in the duration of pharmacological treatment between index and staged procedures)
* Pregnant or breastfeeding women at time of enrolment
* Participation in another trial with an investigational drug or device

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 200 (Estimated)
Dates: Start 2023-07-15 (Actual); Primary Completion 2026-06-15 (Estimated); Study Completion 2027-01-15 (Estimated)

PRIMARY OUTCOMES:
Primary efficacy endpoint | 6 months
  A composite endpoint consisting of all-cause mortality, myocardial infarction, probable and definite Stent Thrombosis and ischemic stroke (the first event that occurs will be counted for this composite endpoint)
Primary safety endpoint | 6 months
  Composite endpint consisting of major or clinically relevant non-major bleeding (BARC type 2, 3 or 5 bleeding)

SECONDARY OUTCOMES:
Mortality | 3 and 6 months
  all-cause mortality
Myocardial infarction | 3 and 6 months
  Myocardial infarction
Stent thrombosis | 3 and 6 months
  Probable and definite Stent Thrombosis
Ischemic stroke | 3 and 6 months
  ischemic stroke
Major bleeding | 3 and 6 months
  BARC 3 or 5 bleeding
Major bleeding | 3 and 6 months
  BARC 3 bleeding
Clinically relevant non-major bleeding | 3 and 6 months
  BARC 2 bleeding

CONTACTS AND LOCATIONS:
Overall Officials: Ashley Verburg, MD, Study Director — St. Antonius Hospital
Locations (1):
- St. Antonius Hospital, Nieuwegein, Utrecht, Netherlands

IPD SHARING:
Plan to Share IPD: No